CLINICAL TRIAL: NCT05772845
Title: A Controlled Evaluation of Abstinence-Induced Withdrawal and Motivation to Vape/Smoke Among Daily ENDS Users Vs. Cigarette Smokers
Brief Title: Vaping and Smoking Withdrawal Project
Acronym: VASP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Roswell Park Cancer Institute (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Larry Hawk, Ph.D., Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00006122; R01DA054276 (NIH)
Record Dates: First submitted 2023-02-16; First posted 2023-03-16 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Acute Abstinence from Cigarettes Vs E-cigarettes (ENDS)
MeSH Terms: interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: All participants will complete two visits, one following 24-hour abstinence, the other while smoking/vaping as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Daily Users of ENDS (Other): Participants who use nicotine-containing ENDS daily or near-daily but who do NOT smoke combustible cigarettes daily or near-daily.
  Interventions: Behavioral: Acute (24-hour) abstinence; Behavioral: Ad libitum smoking/vaping
- Daily Users of Combustible Cigarettes (Other): Participants who smoke combustible cigarettes daily or near-daily but do NOT use nicotine-containing ENDS daily or near-daily.
  Interventions: Behavioral: Acute (24-hour) abstinence; Behavioral: Ad libitum smoking/vaping
- Daily Dual Users of ENDS and Combustible Cigarettes (Other): Participants who both use nicotine-containing ENDS and combustible cigarettes daily or near-daily
  Interventions: Behavioral: Acute (24-hour) abstinence; Behavioral: Ad libitum smoking/vaping

INTERVENTIONS:
Behavioral: Acute (24-hour) abstinence — Participants will be asked to abstain from all tobacco/nicotine for 24 hours prior to the visit
Behavioral: Ad libitum smoking/vaping — Participants will be asked to smoke/vape as usual during the 24 hours prior to the visit

SUMMARY:
The proposed research, which will systematically and comprehensively characterize the withdrawal among daily vapers compared to daily smokers of combustible cigarettes, filling critical gaps in the understanding of electronic nicotine delivery systems (ENDS) dependence/abuse liability and contributing to the development of therapies for tobacco/nicotine use, the leading preventable cause of death in the US.

DETAILED DESCRIPTION:
Withdrawal is a key, multi-faceted component of tobacco/nicotine dependence. Because withdrawal symptoms are theorized to drive relapse, facets of withdrawal (e.g., craving, negative affect) are the targets of most current and emerging treatments. Despite the central importance of withdrawal, and a voluminous literature on withdrawal from combustible cigarette smoking, little is known about withdrawal from electronic nicotine delivery systems (ENDS). To overcome critical barriers to progress in the field, the first-ever prospective, controlled comparison of abstinence-induced withdrawal between ENDS vapers and cigarette smokers is proposed. Participants will be 160 established daily vapers (including former smokers and dual users who smoke occasionally), 160 established daily smokers (including former vapers and dual users who vape occasionally), and (for exploratory comparisons) 50 established daily dual users, who smoke and vape daily. Participants will complete two 4-hour lab visits; the order of the ad lib use visit and the abstinent visit (which follows 24 hours of abstinence) will be randomized across participants. To advance knowledge of ENDS withdrawal, state-of-the-science, multi-measure, multi-method assessments of key withdrawal facets (negative affect, craving, difficulty concentrating, restlessness, sleep, and appetite, as well as anhedonia/positive affect and somatic effects) will be employed. For each facet, the hypothesis that withdrawal magnitude is lower among vapers compared to smokers will be tested. To inform theory and intervention development, the behavioral significance of ENDS withdrawal will also be evaluated, testing the hypotheses that abstinence will increase the motivation to vape/smoke and this group difference will be accounted for (mediated) by vaper/smoker differences in one or more withdrawal facets. Exploratory analyses will examine whether group differences in withdrawal are accounted for (mediate) by differential nicotine exposure, explore the role of individual differences (e.g., sex, rate of nicotine metabolism, expectancies), and examine differences among sub-groups of vapers. The impact of this much-needed, detailed characterization of withdrawal from ENDS is enhanced by the inclusion of a comparator of great public health significance, cigarette smoking. In addition, by characterizing the specific withdrawal facets that drive motivation to vape/smoke, the proposed work will identify promising intervention targets for subsequent treatment development efforts.

ELIGIBILITY:
Inclusion Criteria:

* 6+ months of daily/near-daily nicotine vaping and/or cigarette smoking (to yield 160 vapers, 160 smokers, 50 dual users)
* 200+ ng/mL cotinine on a commercially-available quick screen

Current Exclusion Criteria:

* intention to quit daily/near-daily vaping/smoking in the next month
* current (2+ days out of the past 7) use of pipe tobacco, hookah/shisha, smokeless tobacco, dissolvable tobacco, nicotine pouches. For vaping group only, current (2+ days out of past 7) use of cigars, cigarillos, or filtered cigars that are filled with tobacco or a mix of tobacco and marijuana
* current use of any smoking cessation medication
* current severe substance dependence other than tobacco/nicotine (including cannabis; NIDA Modified ASSIST of 27+)
* current (past 2 weeks) suicidal ideation with intent and/or plan
* current antipsychotic medications or lifetime history of schizophrenia or bipolar disorder
* pregnancy (intake urine screen)

Original Exclusion Criteria that have been modified or eliminated:

* >1 use in past month of tobacco/nicotine products other than ENDS and combustible cigarettes (modified 5/19/25 - see current exclusion criteria)
* alcohol: AUDIT > 15 for males and >13 for females (eliminated 7/25/23)
* current major depression (PHQ-9>11) (eliminated 7/25/23)
* suicide risk (answer to question #9 on PHQ-9 is anything other than "Not at all") (modified 11/17/23 - see current exclusion criteria)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 370 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Wisconsin Smoking Withdrawal Scale - anger 0.5 | 0.5 hours
  anger subscale score
Wisconsin Smoking Withdrawal Scale - anger 2.5 | 2.5 hours
  anger subscale score
Wisconsin Smoking Withdrawal Scale - anx 0.5 | 0.5 hours
  anxiety subscale score
Wisconsin Smoking Withdrawal Scale - anx 2.5 | 2.5 hours
  anxiety subscale score
Wisconsin Smoking Withdrawal Scale - sad 0.5 | 0.5 hours
  sadness subscale score
Wisconsin Smoking Withdrawal Scale - sad 2.5 | 2.5 hours
  sadness subscale score
Wisconsin Smoking Withdrawal Scale - conc 0.5 | 0.5 hours
  difficulty concentrating subscale score
Wisconsin Smoking Withdrawal Scale - conc 2.5 | 2.5 hours
  difficulty concentrating subscale score
Wisconsin Smoking Withdrawal Scale - sleep 0.5 | 0.5 hours
  sleep subscale score
Wisconsin Smoking Withdrawal Scale - sleep 2.5 | 2.5 hours
  sleep subscale score
Wisconsin Smoking Withdrawal Scale - appetite 0.5 | 0.5 hours
  appetite subscale score
Wisconsin Smoking Withdrawal Scale - appetite 2.5 | 2.5 hours
  appetite subscale score
Mood and Physical Symptoms Scale - 0.5 | 0.5 hours
  single-item indicators of withdrawal facets
Mood and Physical Symptoms Scale - 2.5 | 2.5 hours
  single-item indicators of withdrawal facets
Minnesota Nicotine Withdrawal Scale - 0.5 | 0.5 hours
  17-item version with indicators of various withdrawal facets
Minnesota Nicotine Withdrawal Scale - 2.5 | 2.5 hours
  17-item version with indicators of various withdrawal facets
Positive and Negative Affect Scale - PA 0.5 | 0.5 hours
  positive affect subscale score
Positive and Negative Affect Scale - PA 2.5 | 2.5 hours
  positive affect subscale score
Positive and Negative Affect Scale - NA 0.5 | 0.5 hours
  negative affect subscale score
Positive and Negative Affect Scale - NA 2.5 | 2.5 hours
  negative affect subscale score
Snaith-Hamilton Pleasure Scale 0.5 | 0.5 hours
  total score
Snaith-Hamilton Pleasure Scale 2.5 | 2.5 hours
  total score
Questionnaire on Vaping Craving 0.5 | 0.5 hours
  total craving score
Questionnaire on Vaping Craving 2.5 | 2.5 hours
  total craving score
Questionnaire on Smoking Urges - Brief 0.5 | 0.5 hours
  total craving score
Questionnaire on Smoking Urges - Brief 2.5 | 2.5 hours
  total craving score
PhenX Toolkit Insomnia Severity Index 0.5 | 0.5 hours
  7-item scale (but item #5 is omitted because of the short time-frame), total score impairment and interference with daily functioning
PhenX Toolkit Insomnia Severity Index 2.5 | 2.5 hours
  7-item scale (but item #5 is omitted because of the short time-frame), total score impairment and interference with daily functioning
Restlessness ratings 0.5 | 0.5 hours
  3-item scale
Restlessness ratings 2.5 | 2.5 hours
  3-item scale
Restlessness and Agitation Questionnaire - Modified 0.5 | 0.5 hours
  total score on subset of behavioral indicators
Restlessness and Agitation Questionnaire - Modified 2.5 | 2.5 hours
  total score on subset of behavioral indicators
Identical Pair Continuous Performance Task | ~2 hours
  Sustained attention, or vigilance, is the ability to maintain alertness to detect infrequent target stimuli during a long, monotonous task (e.g., Mackworth, 1948). We will use a version of the identical-pairs continuous performance task (Cornblatt et al., 1988) in which participants attend to a series of 800 4-digit numbers on a computer monitor (100-ms stimulus duration; 1500-ms ISI).
  Participants are asked to press the keyboard space bar only when the stimulus is identical to the immediately preceding stimulus (10% targets; Cooper et al., 2020; Rhodes & Hawk, 2016).
  Percent correct hits (target detections) is the primary outcome.
n-back working memory task | ~2 hours
  The n-back task (e.g., Strand et al., 2012; Rhodes & Hawk, 2016) requires indicating whether each stimulus in a rapidly presented series matches the location of the stimulus presented n stimuli before (e.g., n=0,1,2). Stimuli are small grey circles (100 ms; 30% targets). The focus here is on conditions that place marked demands on the "central executive" by requiring ongoing mental manipulation (i.e., n=2; see Baddeley, 2003). Brief practice with a 1-back and 2-back will be followed by 2 100-trial blocks of the 2-back. Accuracy is the primary outcome.
Stop signal reaction time task | ~2 hours
  We will employ the stop-signal paradigm (Logan et al., 1984), which provides a relatively pure index response inhibition (e.g., Nigg, 2001). In our typical task (e.g., Hawk et al., 2018; Rhodes & Hawk, 2016), participants button press to indicate whether the "go" signal (<-- or -->) is pointing left or right. After a brief "go" practice, the stop signal (100-ms tone) is introduced, and participants complete 3 64-trail bocks during with they are asked to respond as quickly as possible but to not respond on stop signal trials (25% of trials). The stop signal occurs after go signal onset and adjusts dynamically across trials to yield ~50% inhibition (Logan et al., 1997). The primary outcome is stop signal reaction time (SSRT), an estimate of the speed of inhibition.
kcal consumed | 3 hours
  Fat, protein, and carbohydrate calories, and total calories, consumed during the visit.
Hypothetical commodity purchase task - vaping intensity 0.5 | 0.5 hours
  Intensity of demand
Hypothetical commodity purchase task - vaping intensity 2.5 | 2.5 hours
  intensity of demand
Hypothetical commodity purchase task - vaping persistence 0.5 | 0.5 hours
  persistence of demand
Hypothetical commodity purchase task - vaping persistence 2.5 | 2.5 hours
  persistence of demand
Hypothetical commodity purchase task - smoking intensity 0.5 | 0.5 hours
  intensity of demand
Hypothetical commodity purchase task - smoking intensity 0.5 | 2.5 hours
  intensity of demand
Hypothetical commodity purchase task - smoking persistence 0.5 | 0.5 hours
  persistence of demand
Hypothetical commodity purchase task - smoking persistence 2.5 | 2.5 hours
  persistence of demand
Choice Behavior Under Cued Conditions (CBUCC) Task - spend vape | 3 hours
  Spending for vape puffs
Choice Behavior Under Cued Conditions (CBUCC) Task - spend cig | 3 hours
  Spending for cigarette puffs
Choice Behavior Under Cued Conditions (CBUCC) Task - spend water | 3 hours
  Spending for water control
Choice Behavior Under Cued Conditions (CBUCC) Task - crave vape | 3 hours
  Craving for vape puffs
Choice Behavior Under Cued Conditions (CBUCC) Task - crave cig | 3 hours
  Craving for cigarette puffs

SECONDARY OUTCOMES:
modified Cigarette evaluation questionnaire | 3.5 hours
  subjective/sensory aspects of smoking
modified e-Cigarette evaluation questionnaire | 3.5 hours
  subjective/sensory aspects of vaping
Heart rate | assessed at ~30-minute intervals
  Heart rate, in beats per minute
Somatic/side effect checklist | 0.5 hours
  Assesses a range of somatic and psychological symptoms (e.g., headache, fatigue, anxiety)
Somatic/side effect checklist | 2.5 hours
  Assesses a range of somatic and psychological symptoms (e.g., headache, fatigue, anxiety)

OTHER OUTCOMES:
Cotinine | 0.25 hours
  assay cotinine from urine sample collected at the start of each visit in order to assess the degree of compliance with the abstinence manipulation
Expired-air carbon monoxide | 0.25 hours
  biochemical measure related to past 24-hour smoking

CONTACTS AND LOCATIONS:
Overall Officials: Larry Hawk, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to make the full de-identified data set with metadata available through the National Addiction and HIV Data Archive Program (NAHDAP).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared at approximately the same time as the acceptance for publication of the main findings from the final dataset. The dataset will have a permanent digital object identifier and will be available as long as the NAHDAP is available.
Access Criteria: Per NAHDAP